CLINICAL TRIAL: NCT03554226
Title: Agitation and Aggressivity in Alzheimer's Disease Patients: A Cohort Study
Acronym: A3C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Ethypharm (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RC31/14/7163; 2014-A00673-44 (Other: ANSM/ID-RCB)
Record Dates: First submitted 2017-11-05; First posted 2018-06-13 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: Alzheimer Disease
Keywords: agitation; aggressivity
MeSH Terms: conditions — Alzheimer Disease; Psychomotor Agitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AD Patients with NeuroPsychiatric Inventory Clinician (NPI-C) (Experimental): The investigation aims to study the natural evolution of type A / A SPCDs in patients with AD. In this study, patients will receive optimized management based on existing best practice recommendations (HAS Recommendations 2009). It will therefore be a standard care study, since this survey applies the current recommendations on tools for the evaluation of SPCDs and the management of behavioral disorders in Alzheimer's disease (Recommendations HAS 2009).
  Interventions: Behavioral: NeuroPsychiatric Inventory Clinician (NPI-C)

INTERVENTIONS:
Behavioral: NeuroPsychiatric Inventory Clinician (NPI-C) — All scales that will be administered to the patient during this study, (ADL, MMSE, QoL-AD, NPI and CMAI), are the subject of recommendations for the management of patients with AD (HAS 2009, HAS 2011)

SUMMARY:
General Hypothesis: hypothesize that A / A symptoms of AD follow a particular course, influenced by associated factors, and a prospective longitudinal observational study specifically evaluating A / A symptoms in patients with MA, living in an institution and at home, would provide useful data for both clinical practice and research.

Specific Hypothesis: hypothesize that in patients with AD with clinically significant A / A there is a correlation between assessment of A / A severity based on specific scales of A / A and overall impression assessment of clinical improvement or worsening of these symptoms by the clinician.

ELIGIBILITY:
Inclusion Criteria:

1256/5000

* Patient with AD according to NINCDS-ADRDA criteria with or without cerebrovascular component at all stages of the disease.
* Patient with agitation / aggression (A / A) type SPCDs, assessed with a score ≥ 4 of at least 1 of the A / A domains, disinhibition, irritability and / or aberrant motor behavior of the NPI scale, with a score frequency ≥2 during the inclusion visit.
* Participation agreement signed by the patient or, in the event of the patient's incapacity, by his / her legal representative or, as the case may be, by the person of trust or family. The patient's ability to sign informed consent is evaluated by a clinician experienced in the field of dementia.
* Patient with social security

If the patient lives at home:

* Presence of a clearly identified primary caregiver: Person from the entourage of the patient who assumes the main part of the care (at least 2 hours at least 3 times during the week) able to complete the questionnaires and to evaluate the patient.
* Availability and agreement of the carer to accompany the patient during consultations.

If the patient lives in an institution:

• He / she must have been there for at least 2 months before inclusion.

Exclusion Criteria:

745/5000

* Brain pathology (other than AD) that may be the cause of dementia: extensive cerebrovascular disease, Parkinson's disease, Lewy body dementia, frontotemporal dementia, brain trauma.
* A / A secondary to concomitant medications, or to a medical or psychiatric condition
* Concurrent major depressive episode (DSM-IV).
* Psychotic symptoms of delirium type and hallucination clinically significant (score ≥ 4 field delusions and / or hallucinations of the NPI scale).
* Presence of concomitant pathologies preventing participation in the study (testing and / or study visits).
* Concurrent participation in another research that may influence the testing of our study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2014-11-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Severity of A/A with NeuroPsychiatric Inventory Clinician (NPI-C) | Change between enrollment and 12 months
  The severity of the A / A will be evaluated using the scale:
  NeuroPsychiatric Inventory Clinician (NPI-C): combined score of 2 domains agitation and aggression (from Medeiros, 2010).
  The purpose of the NPI-C is to collect information on the presence of neuropsychiatric symptoms in patients with cerebral pathologies.
  The rating of all the behavioral domains of the NPI-C scale (C for Clinician) also makes it possible to measure the scores of the other symptoms.
The clinical relevance of the change observed by the clinician with Alzheimer's Disease Cooperative Study-Clinical Global Impression of Change (ADCS-CGIC) | Change between enrollment and 12 months
  The clinical relevance of the change observed by the clinician will be based on the A / A-specific section of the modified Alzheimer's Disease Cooperative Study-Clinical Global Impression of Change (ADCS-CGIC) (Drye et al, 2012).
  The ADCS-CGIC was developed to evaluate the clinical significance of the evolutions observed in therapeutic trials on Alzheimer's disease, and is based on the measured changes compared to the initial evaluation. The modified version, mADCS-CGIC, evaluates the clinical relevance of a treatment based on the measurement of changes assessed by a clinician. The assessment is performed by a trained clinician at the scale

SECONDARY OUTCOMES:
Cohen-Mansfield Agitation Inventory | Change between enrollment and 12 months
  The original version contains 29 items and contains verbal aggression, physical items and items not related to aggression. The rating of items is done on the occurrence of the frequency of disorders in the previous two weeks on a scale of 0 to 7.
Quality of Life QoL-AD | Change between enrollment and 12 months
  Quality of life for patients and caregivers will be based on the QoL-AD scale at V0, V3, V6 and V12.
  Quantitative variable, therefore this evaluation criterion will be expressed as an average. The passing of the scale lasts approximately 5 minutes. This scale will be evaluated by a TEC : The QOL-AD is administered in interview format to individuals with question the quality of life for Alzheimer's patients

CONTACTS AND LOCATIONS:
Overall Officials: Maria SOTO, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Toulouse University Hospital (CHU de Toulouse), Toulouse, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] De Mauleon A, Delrieu J, Cantet C, Vellas B, Andrieu S, Rosenberg PB, Lyketsos CG, Soto Martin M. Longitudinal Course of Agitation and Aggression in Patients with Alzheimer's Disease in a Cohort Study: Methods, Baseline and Longitudinal Results of the A3C Study. J Prev Alzheimers Dis. 2021;8(2):199-209. doi: 10.14283/jpad.2020.66. PMID 33569568